CLINICAL TRIAL: NCT01359878
Title: Fibrinogen Concentrate as Initial Treatment for Postpartum Haemorrhage - A Randomised Clinically Controlled Trial
Brief Title: Fibrinogen Concentrate as Initial Treatment for Postpartum Haemorrhage: A Randomised Clinically Controlled Trial
Acronym: FIB-PPH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Rigshospitalet, Denmark (Other); Copenhagen University Hospital, Hvidovre (Other); Hillerod Hospital, Denmark (Other); Blood Bank of the Danish capital region (Unknown); Unit for monitoring of Good Clinical Practice Copenhagen University (Unknown); Danish Council for Independent Research (Other); Herlev Hospital (Other); Laerdal Foundation (Other); Aase and Ejnar Danielsens Foundation (Other); The Foundation of 17.12.1981 (Other); Fonden til Lægevidenskabens Fremme (Other); Hans og Nora Buchards Fond (Unknown); Haemonetics Corporation (Industry)
Responsible Party: Principal Investigator, Anne Juul Wikkelsø, MD, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2009-017736-41; 2009-017736-41 (EudraCT Number); 1002168 (Other: The Central Danish National Ethics Comitee); 2612-4233 (Other: The Danish Medicines Agency); 2007-58-0015-00911 (Other: The Danish Data Protection Agency); H-3-2010-004 (Other: The ethical comitee of Capital Region); 2009-315 (Other: The monitoring Unit of Good Clinical Practice, Copenhagen University)
Record Dates: First submitted 2011-05-20; First posted 2011-05-25 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Postpartum Haemorrhage
Keywords: Postpartum haemorrhage; Postpartum bleeding; Postnatal bleeding; Fibrinogen concentrate; Transfusion; Haemostatis; Thrombelastography
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Fibrinogen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fibrinogen Concentrate (Experimental)
  Interventions: Drug: Fibrinogen Concentrate
- Placebo (Placebo Comparator): Isotonic Saline
  Interventions: Drug: Isotonic Saline

INTERVENTIONS:
Drug: Fibrinogen Concentrate — 2 gram intra venous
  Other Names: Haemocomplettan, CSL Behring
  Arms: Fibrinogen Concentrate
Drug: Isotonic Saline — Isotonic saline in equivalent volume - 100 ml
  Arms: Placebo

SUMMARY:
Severe maternal bleeding is a serious complication of birth and causes 125.000 deaths worldwide each year. The investigators aim to investigate if early treatment with fibrinogen concentrate versus saline can reduce the incidence of blood transfusion in women with postpartum haemorrhage.

A low level of fibrinogen has been associated with increased blood loss and transfusion requirements in different clinical settings including obstetrical bleeding. Early up-front treatment with fibrinogen may reduce incidence of transfusion by securing optimal haemostatic capacity in women with postpartum haemorrhage.

The investigators plan to enrol 245 patients on four hospitals in the Capital Region of Denmark during a two year period.

As safety measure the investigators plan to use TEG®/Functional Fibrinogen/Rapid-TEG as haemostatic monitoring of all participants during the trial: Baseline test is taken at inclusion before administration of fibrinogen concentrate/placebo. Further tests are taken immediately after intervention, 4 hours and 24 hours after. Baseline test is blinded to the providers of treatment - the rest is clinically available.

DETAILED DESCRIPTION:
Experimental design Design: We plan to conduct a randomised double-blinded clinically controlled trial: The participants are assigned to either 1) placebo (100 ml of isotonic saline) i.v. or 2) the intervention drug: 2 g of fibrinogen concentrate (Haemocomplettan, CSL Behring) i.v. We intend to use a fixed dose for all patients randomized to the intervention group without prior measurement of the fibrinogen level. This strategy is primarily based on the clinical urgency since the treatment is required to be administered as early as possible.

Materials and duration of study Patients will be included during a two year period at the four largest hospitals in the Capital Region: Rigshospitalet, Hvidovre, Hillerød and Herlev if they fulfil the following eligibility criteria Plan of trial execution In order to secure the ethical aspect "Time for reflection" we will provide all pregnant women who appear in the centres during the trial period with written information on the trial during their midwife evaluation. Only 1,75% of these women are estimated to meet the inclusion criteria postpartum.

Intensive haemostatic monitoring Haemostatic blood samples including thrombelastography (TEG®), functional fibrinogen-assay for TEG®, Rapid-TEG, fibrinogen-level, d-Dimer, INR (international normalized ratio), platelet count and Antithrombin III will be drawn 15 minutes after the intervention is given, 4 hours and 24 hours later. The samples taken after the intervention are fully available for evaluation by the clinicians responsible for the patient. The patient will be observed with blood pressure, pulseoximetry, ECG and possible side effects or re-bleeding will be evaluated.

Follow up The patients will remain hospitalized for a minimum of 24 hours. We will contact all participants by phone six weeks after the intervention. Upon discharge from the hospital, all included patients receive information-material addressing possible late side effects and a contact number.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent from participant.
2. Women who develop PPH defined as bleeding from uterus and/or the birth canal within 24 hours postpartum.
3. Age ≥ 18 years.
4. If vaginal birth: indication of one of the following procedures at the operation theatre with anaesthetic assistance: a) Estimated blood loss ≥ 500 ml and indication of manual removal of placenta or b) Indication of manual exploration of the uterus due to continuous bleeding after the birth of placenta.
5. If birth by Caesarean section: A perioperative blood loss ≥ 1000 ml.

Exclusion Criteria:

1. Patients with known inherited deficiencies of coagulation.
2. Patients in anti-thrombotic treatment prepartum due to increased risk of thrombosis.
3. Patients with a pre-pregnancy weight <45 kg.
4. Patients who refuse to receive blood transfusion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Incidense of transfusion with allogenic blood products | During hospital stay or until 6 weeks postintervention

SECONDARY OUTCOMES:
Severe Postpartum Haemorrhage (PPH) | During hospital stay or until 6 weeks postintervention
  Development of "Severe PPH" defined as: "Decrease of haemoglobin (Hb) of > 2,5 mmol/L, transfusion of at least 4 Red Blood Cell (RBC) units, haemostatic intervention (angiographic embolization, surgical arterial ligation or hysterectomy) or death.
Estimated blood loss | During hospital stay During hospital stay or until 6 weeks postintervention
Total amount of blood transfused | During hospital stay During hospital stay or until 6 weeks postintervention
The development of re-bleeding | Untill follow-up 6 weeks postintervention
  Defined as bleeding reoccuring after primary haemostasis, and requiring surgical procedures or intervention
Hemoglobin level below 3,6 mmol/L | During hospital stay or until 6 weeks postintervention
Side-effects including thromboembolic complications | Untill 6 weeks postintervention
  Safety measures/ Potential known side effects such as: Fever, headache, nausea, vomiting, allergic reactions, anaphylaxis and thrombo-embolic complications (deep venous thrombosis, acute myocardial infarct and lung embolus. All suspected unexpected serious adverse reactions will also be reported in accordance with the Good Clinical Practice (GCP) and the Danish Medicines Agency guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Anne J. Wikkelsoe, MD, Principal Investigator — Department of Anaesthesiology, University Hospital of Herlev, Denmark; Ann M. Møller, MD, DmSc, Study Chair — Department of Anaesthesiology, University Hospital of Herlev, Denmark; Jakob Stensballe, MD, PhD, Study Chair — Blood Bank of Danish Capital Region, Rigshospitalet; Jens Langhoff-Roos, MD, DmSc, Study Chair — Department of Obstetrics, Juliane Marie Centre, Rigshospitalet; Arash Afshari, MD, Study Chair — Department of Anaesthesiology, Juliane Marie Centre, Rigshospitalet, Denmark; Hellen McKinnon Edwards, M.D., Study Chair — Dep. of Anaesthesiology, Herlev
Locations (4):
- Denmark (4):
  - Juliane Marie Centre, Rigshospitalet, Copenhagen, Capital Region
  - University Hospital of Herlev, Herlev, Capital Region
  - University Hospital of Hilleroed, Hilleroed, Capital Region
  - University Hospital of Hvidovre, Hvidovre, Capital Region

REFERENCES:
- [Derived] Wikkelso AJ, Edwards HM, Afshari A, Stensballe J, Langhoff-Roos J, Albrechtsen C, Ekelund K, Hanke G, Secher EL, Sharif HF, Pedersen LM, Troelstrup A, Lauenborg J, Mitchell AU, Fuhrmann L, Svare J, Madsen MG, Bodker B, Moller AM; FIB-PPH trial group. Pre-emptive treatment with fibrinogen concentrate for postpartum haemorrhage: randomized controlled trial. Br J Anaesth. 2015 Apr;114(4):623-33. doi: 10.1093/bja/aeu444. Epub 2015 Jan 13. PMID 25586727
- [Derived] Wikkelsoe AJ, Afshari A, Stensballe J, Langhoff-Roos J, Albrechtsen C, Ekelund K, Hanke G, Sharif HF, Mitchell AU, Svare J, Troelstrup A, Pedersen LM, Lauenborg J, Madsen MG, Bodker B, Moller AM. The FIB-PPH trial: fibrinogen concentrate as initial treatment for postpartum haemorrhage: study protocol for a randomised controlled trial. Trials. 2012 Jul 17;13:110. doi: 10.1186/1745-6215-13-110. PMID 22805300